CLINICAL TRIAL: NCT05195021
Title: The Effect of Different Irrigation and Disinfection Methods on Post-operative Pain in Mandibular Molars With Symptomatic Apical Periodontitis: A Randomized Clinical Trial
Brief Title: The Effect of Different Irrigation and Disinfection Methods on Post-operative Pain (PP)
Acronym: PP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Sema Sönmez Kaplan, Assistant Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BİRUNİ-BAP-2020-01-47
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Post-operative Pain; Apical Periodontitis
Keywords: diode laser; EDDY; post-operative pain; sypmtomatic apical periodontitis
MeSH Terms: conditions — Pain, Postoperative; Periapical Periodontitis | interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (conventional irrigation) (Experimental): After finishing the mechanical instrumentation, each root canal was irrigated with 5 ml of 5.25% NaOCl using a 31-gauge needle positioned 2 mm shorter than the WL. To remove the smear layer, 5 ml of 17% ethylenediaminetetraacetic acid (EDTA) was used in each canal for 1 minute, and 5 ml of saline was then administered to neutralize all the residues.
  Interventions: Device: Conventional irrigation
- Group 2 (EDDY) (Experimental): In group 2, 1 ml of 5.25% NaOCl was agitated for 20 seconds three times with the EDDY tip positioned 2 mm shorter than the WL. The root canals were then irrigated with 2 ml of 5.25% NaOCl again. Subsequently, the EDDY tip was activated with short pumping movements, and 2 ml of 17% EDTA was activated for 30 seconds, as described above. The final irrigation followed the same procedures as in group 1.
  Interventions: Device: EDDY; Device: Conventional irrigation
- Group 3 (conventional irrigation and laser irradiation) (Experimental): In group 3, final irrigation followed the same procedures as in group 1 and group 2. During the laser therapy, both the operator and the patient wore eyewear for protection. Laser irradiation was performed using a 980-nm diode laser (Medency Primo 10 W Diode Laser; Vicenza, Italy), coupled with optical fibre (200 µm). The settings were as follows: average power of 1.2 W with a low frequency of 50 Hz and energy of 12 J (each cycle) in pulsed mode, irradiation for 10 seconds, followed by a 10 second pause, which constituted one cycle. This cycle was applied four times to each root canal. The optical fibre tip was located at the WL. The root canals were then slowly (at a speed of 2 mm/s) irradiated from the apical to the coronal portion using a continuous helicoidal movement, with optical fibre tip contacting the root canal walls in one cycle for each power.
  Interventions: Device: Diode Laser device; Device: Conventional irrigation
- Group 4 (EDDY and laser irradiation) (Experimental): In this group, after agitation using the EDDY (VDW) system was performed using the same procedures as in group 3, final irrigation and laser irradiation were done as in group 2.
  Interventions: Device: EDDY; Device: Diode Laser device; Device: Conventional irrigation

INTERVENTIONS:
Device: EDDY — EDDY (VDW) sonic irrigation activation system
  Other Names: EDDY (VDW, Munich, Germany)
  Arms: Group 2 (EDDY); Group 4 (EDDY and laser irradiation)
Device: Diode Laser device — 980-nm diode laser device
  Other Names: Medency Primo 10 W Diode Laser, Vicenza, Italy
  Arms: Group 3 (conventional irrigation and laser irradiation); Group 4 (EDDY and laser irradiation)
Device: Conventional irrigation — Conventional root canal irrigation with 31-guage side port needle
  Other Names: 31-guage side port needle (NaviTip; Ultradent, South Jordan, UT)

SUMMARY:
Aim: The aim of this study was to examine post-operative pain (PP) severity after conventional irrigation and sonic activation methods, with and without laser disinfection in mandibular molar teeth diagnosed with symptomatic apical periodontitis.

Methods: In total, 80 patients with symptomatic apical periodontitis were included in this randomized clinical study. There were four different irrigation and disinfection groups. In group 1, conventional irrigation only was applied. In group 2, EDDY (VDW, Munich, Germany), a sonic irrigation activation system, was applied. In groups 3 and 4, irradiation with a 980-nm diode laser was performed, following irrigation with the conventional method (needle irrigation) and EDDY (VDW) irrigation system, respectively. PP was assessed using a visual analogue scale (VAS). The patients were instructed to record their PP using this scale 8, 24, 48 hours and 7 days post-procedure, in addition to their analgesic intake. A chi-square test, Fisher's exact chi-square test and Fisher-Freeman-Halton exact test were used to assess qualitative data. Inter-group and intra-group parameters were assessed using the Kruskal-Wallis test and Wilcoxon's test at a significance level of p < 0.05 (for both).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult patients aged between 18 and 65 years
2. Moderate to severe pain (4-10) according to a visual analogue scale (VAS)
3. Mandibular molar teeth diagnosed with symptomatic apical periodontitis (a painful response during mastication and/or percussion or palpation)

Exclusion Criteria:

1. Pregnancy or lactation
2. Taking analgesics or anti-inflammatory drugs 12 hours before the treatment
3. Taking antibiotics in the month prior to the treatment
4. Teeth with calcified root canals, greater than grade I mobility and a 4 mm pocket depth, non-restorable damage, occlusal trauma and previous root canal treatment or an open apex
5. Allergy to articaine or non-steroid anti-inflammatory drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | 7 days
  Post-operative pain levels in each group were assessed by visual analog scale (VAS) The pain levels were evaluated at 8, 24, 48 hours and 7 days post-procedure
Anaglesic intake | 7 days
  After the operation nalgesic intake and time intervals were recorded

CONTACTS AND LOCATIONS:
Overall Officials: Sema Sönmez Kaplan, DDS, PhD, Principal Investigator — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Not decided which collected IPD or which IPD that underlie results to share in a publication.

REFERENCES:
- [Derived] Kaplan T, Kaplan SS, Sezgin GP. The effect of different irrigation and disinfection methods on post-operative pain in mandibular molars: a randomised clinical trial. BMC Oral Health. 2022 Dec 13;22(1):601. doi: 10.1186/s12903-022-02651-y. PMID 36514017